CLINICAL TRIAL: NCT01577771
Title: Immunogenicity and Reactogenicity of 13-valent Pneumococcal Conjugate Vaccine Among Infants, Toddlers and Children in Bobo-Dioulasso, Burkina Faso: a Phase 4 Randomized Trial
Brief Title: Immunogenicity and Reactogenicity of PCV13 Among Infants and Children in Burkina Faso
Acronym: PCV13-Bobo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Agence de Médecine Préventive, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCV13-Immunogenicity-Bobo; WS779270 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2012-04-05; First posted 2012-04-16 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal conjugate vaccine; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Child (Active Comparator): 1 dose of Prevnar13 at 2 to 4 years of age
  Interventions: Biological: Prevnar13 (manufactured by Pfizer)
- Toddler 1 dose (Experimental): Single dose of Prevnar13 at 12-15 months of age
  Interventions: Biological: Prevnar13 (manufactured by Pfizer)
- Toddler 2 dose (Active Comparator): 2 doses of Prevnar13 2 months apart beginning at 12-15 months of age
  Interventions: Biological: Prevnar13 (manufactured by Pfizer)
- Infants 2+1 (Experimental): Infants receiving Prevnar13 at 6 weeks, 14 weeks and 9 months. Note: This infant immunization schedule is used in many European countries and in South Africa and has been shown to be immunogenic and effective. However, few head-to-head comparisons of the 2+1 and 3+0 schedules have been conducted.
  Interventions: Biological: Prevnar13 (manufactured by Pfizer)
- Infants 3+0 (Active Comparator): Infants receiving Prevnar13 at 6, 10 and 14 weeks
  Interventions: Biological: Prevnar13 (manufactured by Pfizer)

INTERVENTIONS:
Biological: Prevnar13 (manufactured by Pfizer) — Prevnar13 administered IM in the antero-lateral thigh

SUMMARY:
This study aims to evaluate the immunogenicity and reactogenicity of 13-valent pneumococcal conjugate vaccine among infants, toddlers and children in Bobo-Dioulasso, Burkina Faso. Infants will be randomized to receive vaccine at 6, 10, 14 weeks or at 6 weeks, 14 weeks and 9 months of age. Serotype-specific serum IgG, OPA and nasopharyngeal colonization will be assessed at 6 weeks, 18 weeks, 9 months and 10 months of age. Toddlers 12-15 months of age will be randomized to receive either a single dose of PCV13 or 2 doses 2 months apart. Serotype-specific serum IgG and OPA will be measured pre-dose 1 and again 3 months later. Children 2 to 4 years of age will receive a single dose of PCV13 and have IgG and OPA assessments pre-vaccination and 1 month post-vaccination.

The immunogenicity and reactogenicity of PCV13 in the "standard schedule" groups (e.g. 6, 10, 14 weeks for infants and single dose for toddlers) will be compared to that observed in the PCV13 licensure trials. Within each age group the alternative schedule will be compared to the standard schedule in terms of immunogenicity and impact on nasopharyngeal carriage (infants only).

ELIGIBILITY:
Infants inclusion criteria

* Child has birth weight ≥ 2500g
* Child was born at ≥ 37 weeks of pregnancy or judged to be full-term by midwife or birth attendant
* Mother has resided in Burkina Faso for at least 2 years
* Mother has African nationality
* Child will reside in Bobo-Dioulasso urban area for the duration of the study
* Parent or guardian has given informed consent for child's participation

Infants exclusion criteria

* Child was born with a congenital abnormality
* Child has chronic or acute severe illness requiring specialized medical care
* Child has a blood coagulation disorder
* Mother has known HIV infection
* Child is enrolled in another clinical trial
* Child has known allergy to a component of the vaccine
* Child received a pneumococcal vaccine outside the context of the trial
* Child is 53 days of age or older at 6 week visit
* Child weighs <3500g at the 6 week visit
* Blood draw at 6 week visit was unsuccessful after 3 attempts

Toddlers inclusion criteria

* Child is 12 to 15 months of age
* Child has resided in Burkina Faso since birth
* Child has African nationality
* Child will reside in Bobo-Dioulasso urban area for the duration of the study
* Parent or guardian has given informed consent for child's participation

Toddlers exclusion criteria

* Child has visible signs of severe malnutrition
* Child has chronic or acute severe illness requiring specialized medical care
* Child has a blood coagulation disorder
* Child has known HIV infection
* Child is enrolled in another clinical trial
* Child has known allergy to a component of the vaccine
* Child received a pneumococcal vaccine outside the context of the trial
* Child's weight at first vaccination visit is lower than the 5th percentile of Burkinabe children (8.0 to 8.7 kg according to age)
* Blood draw at first vaccination visit was unsuccessful after 3 attempts

Children inclusion criteria

* Child is 2 to 4 years of age
* Child has resided in Burkina Faso since birth
* Child has African nationality
* Child will reside in Bobo-Dioulasso urban area for the duration of the study
* Parent or guardian has given informed consent for child's participation

Children exclusion criteria

* Child has visible signs of severe malnutrition
* Child has chronic or acute severe illness requiring specialized medical care
* Child has a blood coagulation disorder
* Child has known HIV infection
* Child is enrolled in another clinical trial
* Child has known allergy to a component of the vaccine
* Child received a pneumococcal vaccine outside the context of the trial
* Child's weight at first vaccination visit is lower than the 5th percentile of Burkinabe children
* Blood draw at first vaccination visit was unsuccessful after 3 attempts

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 663 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Serotype-specific pneumococcal serum IgG | 18 weeks for infants
  Primary outcome in other age groups is:
  * 3 months post-dose 1 (toddlers)
  * 1 month post-vaccination (children)

SECONDARY OUTCOMES:
Serotype-specific pneumococcal serum OPA | 18 weeks, 9 months and 10 months (infants), 3 months post-dose 1 (toddlers), 1 month post-vaccination (children)
Vaccine-type and non-vaccine type pneumococcal nasopharyngeal carriage | 18 weeks, 9 months and 10 months (infants)
Adverse events following immunization | 1 and 3 days after each dose of vaccine (active surveillance), up to 28 days post-vaccination (passive surveillance)
Serotype-specific serum IgG | in infants, at 9 months and 10 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bosco Ouedrogo, MD PhD, Principal Investigator — Centre Muraz
Locations (4):
- Burkina Faso (4):
  - CSPS Accart-Ville, Bobo-Dioulasso, Region Des Hauts Bassins
  - Centre Muraz, Bobo-Dioulasso, Region Des Hauts-Bassins
  - CSPS Farakan, Bobo-Dioulasso, Region Des Hauts-Bassins
  - CSPS Guimbi, Bobo-Dioulasso, Region Des Hauts-Bassins